CLINICAL TRIAL: NCT01134640
Title: A Post-Marketing Surveillance Study On Erbitux® (Cetuximab) In Patients With Metastatic Colorectal Cancer Refractory To Irinotecan Containing Treatment
Status: Completed | Type: Observational
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Other Study IDs: ESST
Record Dates: First submitted 2010-05-17; First posted 2010-06-02 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2014-05

CONDITIONS: Metastatic Colorectal Cancer
Keywords: metastatic colorectal cancer; mCRC; post marketing surveillance; Erbitux; Cetuximab; KRAS
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
A post marketing surveillance, prospective study to collect safety information from 250 subjects with epidermal growth factor receptor (EGFR) expressing, KRAS wild-type metastatic colorectal cancer treated with Erbitux as final evaluable cases.

ELIGIBILITY:
Inclusion Criteria:

* EGFR expressing, KRAS wild-type subjects with metastatic colorectal cancer, who are indicated for Erbitux treatment according to the nationally authorized label (in combination with irinotecan, metastatic colorectal cancer after failure of irinotecan-including cytotoxic therapy)

Exclusion Criteria:

* Subjects who are not eligible for Erbitux treatment according to the indication in national label; or with hypersensitivity reactions (grade 3 or 4) to Erbitux

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: EGFR expressing, KRAS wild-type subjects with metastatic colorectal cancer, who are indicated for Erbitux treatment according to the nationally authorized label (in combination with irinotecan, metastatic colorectal cancer after failure of irinotecan-including cytotoxic therapy)
Sampling Method: Non-Probability Sample
Enrollment: 286 (Actual)
Dates: Start 2008-01; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Safety and toxicity of Erbitux in clinical practice | Till 28 days after last dose of Erbitux
  To obtain safety information on the use of Erbitux in subjects with metastatic colorectal cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Jade Lien, Study Director — Merck Ltd., Taiwan
Locations (15):
- Taiwan (15):
  - Chang Gung Medical Foundation, Chiayi City
  - Chiayi Christian Hospital, Chiayi City
  - Buddhist Tzu Chi General Hospital, Hualien City
  - Chang Gung Medical Foundation, Kaohsiung City
  - Chang Gung Medical Foundation, Keelung
  - Chang Gung Medical Foundation, Linkou District
  - Chung Shan Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - Chi Mei Medical Center, Liou Ying, Tainan
  - Chi Mei Medical Center, Yongkang, Tainan
  - National Cheng Kung University Hospital, Tainan
  - Tainan Municipal Hospital, Tainan
  - Buddhist Tzu Chi General Hospital, Taipei
  - Mackay Memorial Hospital, Taipei
  - Shin Kong Wu Ho-Su Memorial Hospital, Taipei